CLINICAL TRIAL: NCT06325748
Title: SENTI-202-101: A Phase 1, Multicenter, Open-Label Study of SENTI-202, a Selective Off-the-Shelf Logic Gated CAR NK Cell Therapy, in Subjects With CD33 and/or FLT3 Expressing Malignancies
Brief Title: SENTI-202: Off-the-shelf Logic Gated CAR NK Cell Therapy in Adults With CD33 and/or FLT3 Blood Cancers Including AML/MDS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Senti Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENTI-202-101
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: AML/MDS; CD33 Expressing Hematological Malignancies; FLT3 Expressing Hematological Malignancies
Keywords: SENTI-202; CAR NK; natural killer cell; CD33; FLT3; allogeneic; logic gate; relapsed/refractory AML; relapsed/refractory MDS; inhibitory CAR; activating CAR; NOT logic gate; IL15; interleukin 15; cell therapy; off-the-shelf; leukemic stem cells; blastic plasmacytoid dendritic cell neoplasm (BPDCN); multiple myeloma (MM); mixed phenotype acute leukemia (MPAL); endomucin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Blastic Plasmacytoid Dendritic Cell Neoplasm; Multiple Myeloma; Leukemia, Biphenotypic, Acute | interventions — fludarabine; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SENTI-202 CAR NK cell therapy (Experimental): Part 1 Dose Finding: Sequential cohorts will receive doses of SENTI-202 using a modified 3+3 study design to determine the recommended phase 2 dose (RP2D). The starting dose will be 1 billion cells. Other doses may be explored depending on study data.
  Part 2 Cohort Expansion: After determination of the RP2D, additional subjects will be enrolled in disease-specific expansion cohorts at that dose to further explore safety, biodynamics, and anti-cancer activity of SENTI-202
  Interventions: Biological: SENTI-202

INTERVENTIONS:
Biological: SENTI-202 — SENTI-202 is an investigational off-the-shelf CAR NK cell therapy designed to selectively target and eliminate CD33 and/or FLT3 expressing hematological malignancies while sparing healthy cells using a NOT logic gate.
  SENTI-202 is administered in either a 3 dose regimen (Schedule 1: Days 0, 7, 14) or a 5 dose regimen (Schedule 2: Days 0, 3, 7, 10, 14) of a 28-day treatment cycle following a lymphodepletion conditioning regimen of fludarabine and cytarabine (flu/Ara-C). Subjects will receive a minimum of 1 and maximum of 3 treatment cycles to achieve optimal response with the optionality of an additional consolidation cycle thereafter. Additional dosing schedules may be explored depending on study data.
  Other Names: Fludarabine; Cytarabine (ara-C)

SUMMARY:
This is an open-label study of the safety, biodynamics, and anti-cancer activity of SENTI-202 (an off-the-shelf logic gated CAR NK cell therapy) in patients with CD33 and/or FLT3 expressing blood cancers, including AML and MDS.

DETAILED DESCRIPTION:
This is a dose-finding study of SENTI-202, comprised of an initial dose finding using a modified "3+3" study design to determine the maximum tolerated dose (MTD) and/or recommended phase two dose (RP2D) of SENTI-202 when administered after lymphodepleting chemotherapy (Part 1) followed by disease-specific expansion cohorts at the RP2D (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD33 and/or FLT3 expressing malignancies, including:

  * Relapsed refractory acute myeloid leukemia (AML) with morphologic relapse as defined by ≥5% bone marrow blasts who have received at least 1 prior line, but no more than 3 prior lines of standard anti-AML therapy. Subjects with FLT3-mutated or IDH ½-mutated disease must have received at least one prior targeted therapy.
  * Relapsed refractory myelodysplastic syndrome (MDS) with increased blasts who have received at least 1 prior line, but no more than 2 prior lines of anti-MDS therapy
  * Other hematological malignancies who have received at least 1 prior line of standard of care for the respective disease
  * Documentation of CD33 expression (or FLT3 expression if available) by individual institutional standard of care
* ECOG performance score of 0-1
* Adequate organ function including platelet count >20x109/L (platelet transfusion is permitted)
* Adequate recovery from toxicities from previous cancer treatments, as described in the study protocol
* Willing and able to provide written informed consent

Exclusion Criteria:

* White blood cell (WBC) count of ≥20×109/L or circulating blasts ≥10×109/L or rapidly progressive/hyperproliferative disease
* Acute promyelocytic leukemia with t(15;17) (q22;q12) or abnormal promyelocytic leukemia/retinoic acid receptor alpha (APML-RARA)
* MDS with fibrosis (MDS-f) or known prior history of constitutional conditions/syndromes with chemo-responsive AML
* Evidence of leukemic meningitis or known active central nervous system disease
* Presence of extra-medullary disease or myeloid sarcoma alone with no morphologic hematologic relapse
* Prior use of certain anti-cancer therapies and/or use within a certain number of days prior to SENTI-202 study treatment, as described in the study protocol
* Hematopoietic cell transplantation (HCT) less than 100 days prior to the first dose of SENTI-202
* Prior NK cell or CAR T cell therapy at any time
* Prior donor lymphocyte infusion (DLI), except if after HCT for MRD+ disease
* Medical conditions or medications prohibited by the study protocol
* Pregnant or breastfeeding female

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability for dose determination of SENTI-202 | At the end of each treatment cycle (each cycle is 28 days) and through study completion, up to 2 years
  Incidence, type, frequency, and severity of adverse events and dose limiting toxicities will be assessed to determine the maximum tolerated dose and/or recommended phase 2 dose and dosing regimen
For subjects enrolled in the Dose Expansion Cohort(s): Anti-cancer activity of SENTI-202 | Through study completion, up to 2 years
  The response rate to SENTI-202 will be measured using clinical measures of benefit as defined by standard consensus criteria for the respective disease

SECONDARY OUTCOMES:
For subjects enrolled in the Dose Finding Cohorts: Anti-cancer activity of SENTI-202 | Through study completion, up to 2 years
  The response rate to SENTI-202 will be measured using clinical measures of benefit as defined by standard consensus criteria for the respective disease
Pharmacokinetic (PK) and pharmacodynamic (PDn) profile of SENTI-202 | Through study completion, up to 2 years
  Levels of circulating SENTI-202 and peripheral cytokine levels will be measured to assess the PK/PDn profile of SENTI-202
Host immune response to SENTI-202 | Through study completion, up to 2 years
  Anti-SENTI-202 immune response and RCR will be measured in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle Emery, MD, Study Director — Senti Biosciences, Medical Director
Locations (8):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare, San Antonio, Texas
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Peter MacCallum Cancer Center, Melbourne, Victoria